CLINICAL TRIAL: NCT06364514
Title: PICNIC Study - PatIent Centered aNtIbiotic Courses in Children With Medical Complexity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Kathleen Snow, Instructor, Pediatrics, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00047313
Record Dates: First submitted 2024-04-03; First posted 2024-04-15 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Patients will be started on antibiotics for treatment of pneumonia per usual care by their medical provider team. The research team will monitor enrolled patients daily for markers of their clinical status (caregiver assessment of respiratory status, supplemental oxygen/respiratory support, presence of fever). Once the patient has been "clinically stable" x48 hours, antibiotics will be discontinued.
  Interventions: Other: Clinical Stability Assessment

INTERVENTIONS:
Other: Clinical Stability Assessment — Base total days of antibiotics on clinical stability vs utilizing predetermined total days of antibiotics

SUMMARY:
To determine if clinicians can safely reduce antibiotic exposure in children with medical complexity (CMC) who are diagnosed with pneumonia by implementing an intervention that bases total antibiotic duration on an individual's clinical stability.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the Complex Care Service at Boston Children's Hospital with a provider diagnosis of pneumonia
* Started on antibiotics by the provider team
* Ages 2-25 years old

Exclusion Criteria:

* Patients initially admitted to the intermediate care unit or ICU due to increased respiratory support needs

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible patients who consent to participate in the intervention | 48 hours
  Caregiver and medical provider acceptability
Rate of persistent and worsening respiratory symptoms measured by patient's clinical status; the rate of emergency department revisit or hospital readmission within 1 week of antibiotic discontinuation | 1 week
  Patient Safety Outcomes

SECONDARY OUTCOMES:
Median days of antibiotics received for patients in the intervention group as well as from historical control group | 30 days
  Pneumonia antibiotic duration

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No